CLINICAL TRIAL: NCT00790270
Title: Comparison of Ibuprofen, Cyclobenzaprine, or Both for Acute Cervical Strain: A Randomized Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Adam Singer, MD, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SB2003-1234
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Results first posted 2012-11-21 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-10

CONDITIONS: Cervical Strain
Keywords: Cervical strain; whiplash; ibuprofen; cyclobenzaprine
MeSH Terms: conditions — Whiplash Injuries | interventions — cyclobenzaprine; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cyclobenzaprine (Active Comparator)
  Interventions: Drug: Cyclobenzaprine
- Ibuprofen (Active Comparator)
  Interventions: Drug: Ibuprofen
- Ibuprophen plus Cyclobenzaprine (Experimental)
  Interventions: Drug: Ibuprofen plus Cyclobenzaprine

INTERVENTIONS:
Drug: Cyclobenzaprine — 5 mg orally every 8 hours as needed
  Other Names: flexeril
  Arms: Cyclobenzaprine
Drug: Ibuprofen — Ibuprofen 400 mg every 8 hours as needed
  Other Names: motrin, advil
  Arms: Ibuprofen
Drug: Ibuprofen plus Cyclobenzaprine — Ibuprofen 400 mg plus cyclobenzaprine 5 mg every 8 hours as needed
  Other Names: motrin or advil with flexeril
  Arms: Ibuprophen plus Cyclobenzaprine

SUMMARY:
The purpose of this study is to see whether the combination of a muscle relaxant and anti-inflammatory drug is more effective at relieving pain in patients with neck strains or whiplash than either of the two medications alone.

DETAILED DESCRIPTION:
Muscle relaxants have been used extensively for neck and back pain since muscle spasm is thought to play a role in the cycle of pain and spasm. However, prior studies have conflicting results regarding their additive effect when given in addition to analgesics such as the NSAIDs. Because they have the potential to lead to adverse events their efficacy should be clearly demonstrated before their routine use.

ELIGIBILITY:
Inclusion Criteria:

* neck pain within 24 hours of injury

Exclusion Criteria:

* Children, allergy or contraindication to any of the study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2003-01; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: adam singer, md, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cyclobenzaprine | Ibuprofen | Ibuprophen Plus Cyclobenzaprine
Started | 21 | 20 | 20
Completed | 21 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyclobenzaprine | Ibuprofen | Ibuprophen Plus Cyclobenzaprine | Total
Number analyzed (Participants) | 21 | 20 | 20 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 20 | 20 | 61
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 36 (13) | 32 (10) | 32 (10) | 33 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 9 | 34
  Male | 7 | 9 | 11 | 27
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 20 | 61

OUTCOME MEASURES:

1. Primary Outcome: Pain
Time Frame: Daily for 1 week
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: mm on visual analog scale

2. Secondary Outcome: Time to Resumption of Work
Time Frame: 1 week
Reporting Status: Not Posted

3. Primary Outcome: Use of Rescue Medications
Description: the number of patients taking additional rescue medications beyond the study meds
Time Frame: 24 hours
Population: number of patients using additionl anlagesics on the day following enrollment
Measure: Number; unit: participants
Arm/Group | Cyclobenzaprine | Ibuprofen | Ibuprophen Plus Cyclobenzaprine
Number analyzed (Participants) | 21 | 20 | 20
participants | 13 | 9 | 9

4. Secondary Outcome: Resumption of Work or School
Description: number of patients resuming regular activity the day following enrollment.
Time Frame: next day
Measure: Number; unit: participants
Arm/Group | Cyclobenzaprine | Ibuprofen | Ibuprophen Plus Cyclobenzaprine
Number analyzed (Participants) | 21 | 20 | 20
participants | 8 | 14 | 13

ADVERSE EVENTS:
Time Frame: next day
Description: th number of patients reporting an adverse event on the day following enrollment and each additional day for 1 week.
Arm/Group | Cyclobenzaprine | Ibuprofen | Ibuprophen Plus Cyclobenzaprine
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes